CLINICAL TRIAL: NCT01347840
Title: Metabolic Factors of Outcomes From Gastric Bypass Surgery
Acronym: Cassini
Status: Terminated | Type: Observational
Why Stopped: Study was terminated for business reasons.
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: CI-10-0004
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Results first posted 2012-05-21 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-04

CONDITIONS: Obesity
Keywords: Obesity Gastric Bypass Roux en Y
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Subjects: This is a one arm study where all the subjects will receive the same treatment and will not be blinded. No subjects will be assigned to different treatment groups.

SUMMARY:
The objective of this study is to determine whether the metabolic, endocrine and energetic response to short term caloric restriction are factors in weight loss in subjects having gastric bypass (GB) surgery.

ELIGIBILITY:
Inclusion Criteria:

Subjects satisfying the following criteria will be considered the screening population and will be eligible for enrollment in this study:

1. Subject is willing to give consent and comply with evaluation and treatment schedule
2. 18 to 65 years of age (inclusive) on date of signing the ICD
3. Subject is scheduled to have non-revisional GB surgery between 2 weeks to 4 months after signing the ICD
4. Able to read, understand, and follow study procedures as outlined in the ICD.

Exclusion Criteria:

Subjects meeting the following criteria will not be eligible for enrollment:

1. Unable or unwilling to attend follow-up visits and examinations
2. Women who are pregnant, nursing at the time of screening, or planning to become pregnant within one year of the GB surgery
3. Clinically active cardiac, renal, hepatic or GI disorders
4. Screening laboratory tests with any of the following:

   * alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST] ≥ 4 times upper limit of normal (ULN) according to VAMC normal ranges
   * AST:ALT > 2:1 according to VAMC normal ranges
   * Serum Creatinine ≥ 1.5 times ULN according to VAMC normal ranges
   * Blood Urea Nitrogen (BUN) ≥ 1.5 times ULN according to VAMC normal ranges
   * Positive test results for Hepatitis A, B or C
5. Clinically active thyroid or lipid disorders:

   * Thyroid-stimulating hormone (TSH) flagged as critical value (per VAMC lab normal ranges)
   * Triglycerides > 400 mg/dL
6. Anemia:

   * Mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), and mean corpuscular hemoglobin concentration (MCHC) outside normal VAMC range; or
   * Hematocrit < 36%
7. Uncontrolled hypertension which required a medication regimen adjustment during the 3 months prior to screening
8. Currently prescribed or taking atypical antipsychotic medication
9. Currently prescribed or taking chronic, long-term, oral corticosteroid medication
10. Diabetes requiring a drug regimen which includes insulin treatment at the time of screening
11. Unwilling or unable to refrain from having a procedure or surgery which involves the removal of skin tissue which could result in weight loss
12. Any medical condition or finding for which the PI used medical discretion to determine the subject should be excluded; or
13. Participation in any other investigational device or drug study (non survey based trial) during the course of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects having gastric bypass (GB) surgery within 4 months of screening visit.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David D'Alessio, MD, Principal Investigator — Veterans Affairs Medical Center, Cincinnati, OH
Locations (1):
- Veterans Affairs Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Subjects
Started | 1 (1 subject enrolled but withdrew consent)
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Excess Weight Loss
Description: Calculated as the difference between the baseline weight and weight at endpoint divided by the difference between baseline weight and ideal body weight using the medium frame range in the Metropolitan Tables for Life Insurance, 1983 x 100.
Time Frame: 16 months
Measure: Number; unit: percentage of excess weight
Arm/Group | All Subjects
Number analyzed (Participants) | 0

2. Primary Outcome: Resting Energy Expenditure
Description: Energy expended at rest (minimal movement) and during fasting. Resting Energy Expenditure can be expressed per minute or per hour or per day.
Time Frame: 16 months
Measure: Number; unit: units on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 0

3. Primary Outcome: Area Under the Curve of Ghrelin and GLP-1
Description: These variables will measure the combined effects of hormone concentration and duration.
Time Frame: 16 months
Measure: Number; unit: units on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 0

4. Secondary Outcome: Area Under the Curve of Timed Gastrointestinal Hormones (Insulin, GIP, Pancreatic Polypeptide, Peptide YY (PYY), Amylin, Glucagon, Pro-Insulin, C-Peptide)
Description: These variables will measure the combined effects of hormone concentration and duration.
Time Frame: 16 months
Measure: Number; unit: units on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 0

5. Secondary Outcome: Adiponectin and Lectin
Description: These laboratory values will be collected at Visit 3, Visit 5, Visit 6, and Visit 10.
Time Frame: 16 months
Measure: Number; unit: units on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 0

6. Secondary Outcome: Subject Questionnaires
Description: The subscales and total scores as set out in the scoring algorithms for Food Craving Inventory-II and Questionnaire on Craving for Sweet and Rich Foods will be presented.
Time Frame: 16 months
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 0

7. Secondary Outcome: Area Under the Curve of Glucose
Description: This variable will measure the combined effects of glucose concentration and duration.
Time Frame: 16 months
Measure: Number; unit: units on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 0

8. Secondary Outcome: Hemoglobin A1c and Lipid Panel
Description: These laboratory values will be collected at Screening, Visit 8, and Visit 10.
Time Frame: 16 months
Measure: Number; unit: units on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 0

9. Secondary Outcome: Body Mass Index
Description: Will be calculated at Screening, Visit 3, Visit 5, Visit 6, Visit 8, and Visit 10.
Time Frame: 16 Months
Measure: Number; unit: units on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 0

10. Secondary Outcome: Percent Weight Loss
Description: (Weight at Baseline - Weight at Each Visit) divided by the (Weight at Baseline).
Time Frame: 16 Months
Measure: Number; unit: percentage of weight loss
Arm/Group | All Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Trial termination due to business needs. One subject enrolled and withdrew consent. Zero subjects completed study. No subject data analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No